CLINICAL TRIAL: NCT01425931
Title: Gastrointestinal Microcirculation During Cardiopulmonary Bypass
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Arndt-H. Kiessling, Head cardiovascular research, Johann Wolfgang Goethe University Hospital
Other Study IDs: O2C-001AHK
Record Dates: First submitted 2011-08-23; First posted 2011-08-30 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: MeSH Heading Cardiac Surgical Procedures; Tree Number E04.100.376; Tree Number E04.928.220
MeSH Terms: interventions — Heart-Lung Machine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Extracorporeal circulation: all patients were measured by microcirculation device O2C
  Interventions: Procedure: Heart Lung machine

INTERVENTIONS:
Procedure: Heart Lung machine — measurement of microcirculation with O2C device

SUMMARY:
O2C is a diagnostic device for non-invasive determination of oxygen supply in microcirculation of blood perfused tissues. The optical sensor is easy to handle and guarantees reproducible examinations of local oxygen supply of tissues in clinics as well as in research. The examinations are without any strain for your patient.

Determines by use of a glass fibre probe:

Blood Flow in Microcirculation Capillary-Venous Oxygen Saturation Blood Filling of Microvessels Blood Flow Velocity This device makes it possible to supervise the local oxygen supply of organs and tissue.

With it is possible to measure locally the amount of oxygen which is transported into the region of interest and to diagnose local oxygen consumption of an organ. O2C's novelty is monitoring the energetic metabolism of cells by measuring the oxygen uptake with an optical sensor probe. Pathological O2-supply, which can lead to angiogenesis or cell-death and subsequently to organ failure, now can be detected in an early state by use of the new sensor system.

One of these new developed sensors are used to place in rectal position during extracorporeal circulation to determine the microcirculation.

ELIGIBILITY:
Inclusion Criteria:

* Patients on extracorporeal circulation

Exclusion Criteria:

* Haemorrhoidal lesions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac surgery patients with ecc
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Blood Flow in Microcirculation | 3 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Goethe University, Frankfurt am Main, Hesse, Germany